CLINICAL TRIAL: NCT05806944
Title: Evaluation of Active Emotional State on the Efficacy of Transcranial Magnetic Stimulation
Brief Title: Transcranial Magnetic Stimulation for Binge Eating Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Darrin J Lee, MD, PhD, Assistant Professor of Neurological Surgery, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS-21-00791
Record Dates: First submitted 2023-03-15; First posted 2023-04-10 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Binge-Eating Disorder
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Intervention Model Description: double-blinded, pseudorandomized crossover
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group A (Experimental): Patients with BED not undergoing symptom provocation
  Interventions: Device: TMS followed by Sham TMS
- Group B (Experimental): Patients with BED not undergoing symptom provocation
  Interventions: Device: Sham TMS followed by TMS
- Group C (Experimental): Patients with BED undergoing symptom provocation
  Interventions: Device: TMS followed by Sham TMS
- Group D (Experimental): Patients with BED undergoing symptom provocation
  Interventions: Device: Sham TMS followed by TMS

INTERVENTIONS:
Device: TMS followed by Sham TMS — double blinded crossover schedule in which participants will undergo TMS and assessment in one visit, followed by sham-TMS and assessment the next visit.
  Arms: Group A; Group C
Device: Sham TMS followed by TMS — double blinded crossover schedule in which participants will undergo sham TMS and assessment in one visit, followed by TMS and assessment the next visit.
  Arms: Group B; Group D

SUMMARY:
The primary goal of this study is to elucidate the impact of disorder provocation on the efficacy of TMS for the treatment of BED. In order to meet this objective, the investigators propose to evaluate this relationship in using a crossover study. Secondary objectives of this study include determining whether TMS with or without BED symptom provocation has effects in altering neurophysiology as detected by fMRI.

DETAILED DESCRIPTION:
Current literature has demonstrated that transcranial magnetic stimulation (TMS) targeting the dorsolateral prefrontal cortex (DLPFC) has some efficacy in treating binge eating disorder. The investigators believe that TMS may be beneficial in the treatment of binge eating disorder. The purpose of this study is to determine whether TMS has efficacy for binge eating disorder and if symptom provocation affects treatment. This study will be conducted as a pilot study in the Keck Hospital clinics. 32 adult patients with a clinical diagnosis of binge eating disorder will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* English speaking (EPSI and Binge Eating Disorder Scale available only in English)
* Diagnosed with binge eating disorder as defined by the DSM-5 and in treatment for at least 6 months
* Stable doses of medications for at least 6 weeks
* Female subjects of childbearing age must consent to pregnancy tests at the beginning of each treatment session; will be counseled to use barrier methods during the course of this study

Exclusion Criteria:

Contraindications to receiving TMS such as:

1. Aneurysm clips or coils
2. Stents in the neck or brain
3. Deep brain stimulators
4. Electrodes to monitor brain activity
5. Metallic implants in ears and eyes
6. Shrapnel or bullet fragments in or near the head
7. Facial tattoos with metallic or magnetic-sensitive ink
8. Other metal devices or object implanted in or near the head

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The effect of symptom provocation on TMS-mediated changes in the blood-oxygen-level-dependent(BOLD) signal | 33 Days
  BOLD signals measure neural activity indirectly via neurovascular coupling
  Changes in BOLD signals from baseline after TMS +/- symptom provocation will be compared after completion of the crossover study (day 33).
The effect of symptom provocation on TMS-mediated changes in the functional connectivity (FC) within and between pathophysiologically-relevant networks. | 33 Days
  FC measures correlation in activity between different brain regions.
  Changes in FC from baseline after TMS +/- symptom provocation will be compared after completion of the crossover study (day 33).
The effect of symptom provocation on TMS-mediated changes in the behavioral inhibition system (BIS)/behavioral activation system (BAS) scale score | 33 Days
  BIS/BAS scale is a self reported 24 item questionnaire that assesses the BIS, a motivation system for avoiding aversive outcomes, and BAS, a motivation system for approaching goal-oriented outcomes. The total score for BIS scale ranges from 0 to 28 (7 items ranging from 0-4). The total score for BAS ranges from 0 to 52 (13 items ranging from 0-4). Four questions are fillers. Higher score represents greater severity of symptoms.
  Changes in BIS/BAS scale from baseline after TMS+/- symptom provocation will be compared after completion of the crossover study (day 33).
The effect of symptom provocation on TMS-mediated changes in the Eating Disorder Examination - Questionnaire (EDE-Q) | 33 days
  The EDE-Q is a self report questionnaire of ED symptomatology over the preceding 28 days, that encompasses behavioral and attitudinal symptoms across four domains - dietary restraint, eating concern, shape concern, and weight concern. The subscores are calculated as follows:
  Restraint = (Item 1 + Item 2 + Item 3 + Item 4 + Item 5) / 5; Eating Concern = (Item 6 + Item 7 + Item 9 + Item 15 + Item 34) / 5; Weight Concern = (Item 11 + Item 14 + Item 29 + Item 31 + Item 32) / 5; Shape Concern = (Item 10 + Item 11 + Item 12 + Item 13 + Item 30 + Item 33 + Item 35 + Item 36) / 8; Global Score = (Restraint + Eating Concern + Weight Concern + Shape Concern) / 4 Higher score represents greater severity of symptoms.
  Changes in the EDE-Q score from baseline after TMS +/- symptom provocation will be compared after completion of the crossover study (day 33).
The effect of symptom provocation on TMS-mediated changes in the Eating Disorder (ED 15) questionnaire. | 33 days
  The ED 15 questionnaire is a measure of eating disorder symptomatology, designed to measure dynamic, session-by-session fluctuations in ED symptom severity. The overall score ranges from 0-6, as it is calculated as the mean of the scores on all ten items, each ranging from 0-6 on symptom severity. Higher score represents greater severity of symptoms.
  Changes in the ED 15 questionnaire score from baseline after TMS +/- symptom provocation will be compared after completion of the crossover study (day 33).

CONTACTS AND LOCATIONS:
Overall Officials: Darrin J Lee, MD PhD, Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: No